CLINICAL TRIAL: NCT00840632
Title: A Two-Way Crossover, Open-Label, Single-Dose, Fasting, Bioequivalence Study of Trandolapril 4 mg Tablets Versus Mavik® 4 mg Tablets in Normal Healthy Non-Smoking Male and Female Subjects
Brief Title: Trandolapril 4 mg Tablet Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2977
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — trandolapril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trandolapril (Experimental): Trandolapril 4 mg Tablet (test) dosed in first period followed by Mavik® 4 mg Tablet (reference) dosed in second period
  Interventions: Drug: Trandolapril 4 mg Tablets
- Mavik® (Active Comparator): Mavik® 4 mg Tablet (reference) dosed in first period followed by Trandolapril 4 mg Tablet (test) dosed in second period
  Interventions: Drug: Mavik® 4 mg Tablets

INTERVENTIONS:
Drug: Trandolapril 4 mg Tablets — 1 x 4 mg, single-dose fasting
  Arms: Trandolapril
Drug: Mavik® 4 mg Tablets — 1 x 4 mg, single-dose fasting
  Arms: Mavik®

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of trandolapril from a test formulation of Trandolapril 4 mg Tablets versus the reference Mavik® 4 mg Tablets under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria

* Non-smoking male or female with a minimum age of 18 years (i.e. non-smoker or non-tobacco user for at least 90 days prior to pre-study medical screening).
* Body Mass Index (BMI = weight/height2) greater than or equal to 19.0 kg.m2 and less than or equal to 30.0 kg/m2.
* Normal findings in the physical examination, 12-lead ECG and vital signs (blood pressure between 100-140/60-90 mmHg, heart rate between 50-100 beats/min, temperature between 35.8°C and 37.5°C).
* Negative for drugs of abuse, nicotine, hepatitis B-surface antigen, hepatitis C and HIV, and for female subjects, pregnancy (serum β-CG).
* No clinical laboratory values outside of the acceptable range as defined by BCR, unless the Principal Investigator decides they are not clinically significant.
* Female subjects who are surgically sterile for at least six months or post-menopausal for at least one year, or who will avoid pregnancy prior to the study, during the study and up until one month after the end of the study.

Exclusion Criteria

* Known history of hypersensitivity to trandolapril (e.g. Mavik®) other ACE inhibitors such as captopril, benazepril, enalapril, lisinopril, ramipril, quinapril, or cilazapril or angiotensin receptor agonists such as losartan, candesartan, eprosartan, irbesartan, telmisartan, or valsartan.
* Known history or presence of cardiac, pulmonary, gastrointestinal, endocrine, musculoskeletal, neurological, hematological, liver or kidney disease, unless judged not clinically significant by the Principal Investigator or medical designate.
* Known history or presence of food allergies, or any condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness during the last four weeks prior to entry into this study.
* Presence of any significant physical or organ abnormality.
* Any subject with a history of drug abuse.
* Any history or evidence of psychiatric or psychological disease (including depression) unless deemed not clinically significant by the Principal Investigator, or medical designate.
* Use of any prescription medication within 14 days preceding entry into this study.
* Use of over the counter (OTC) medication within seven days preceding entry into this study (except for spermicidal/barrier contraceptive products).
* Female subjects: use of contraceptives (oral, transdermal, implant, Mirena® IUD) within 30 days prior to drug administration or a depot injection of progestogen drug (e.g. Depo-Provera®) within one year prior to drug administration.
* Female subjects: presence of pregnancy or lactation.
* Any subject who has had blood drawn within 56 days preceding this study, taken during the conduct of any clinical study at a facility other than BCR, or within the lockout period specified by a previous study conducted at BCR.
* Participation in a clinical trial with an investigational drug within 30 days preceding this study.
* Any subject who has donated blood within 56 days preceding this study.
* Any subject who has participated as a plasma donor in a plasmapheresis program within seven days preceding this study.
* Significant or recent history of asthma (after 12 years of age).
* Any subject with a recent (less than one year) history of alcohol abuse.
* Known history of frequent headaches or migraines.
* Known history of hereditary or idiopathic angioedema.
* Any history of severe allergic reaction (including drugs, food, insect bites, environmental allergens).
* Intolerance to venipuncture.
* Any clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoine, glucocorticoids, omeprazole,; examples of inhibitors: antidepressant (SSRI), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to administration of the study medication.
* Difficulty swallowing study medication.
* Difficulty fasting or consuming standard meals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-10; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Y Tam, M.D., Principal Investigator — Biovail
Locations (1):
- Biovail Contract Research, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Trandolapril (Test) First: Trandolapril 4 mg Tablet (test) dosed in first period followed by Mavik® 4 mg Tablet (reference) dosed in second period
- Mavik® (Reference) First: Mavik® 4 mg Tablet (reference) dosed in first period followed by Trandolapril 4 mg Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Trandolapril (Test) First | Mavik® (Reference) First
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout
Arm/Group | Trandolapril (Test) First | Mavik® (Reference) First
Started | 20 | 19
Completed | 19 | 18
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Second Intervention
Arm/Group | Trandolapril (Test) First | Mavik® (Reference) First
Started | 19 | 18
Completed | 19 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trandolapril (Test) First | Mavik® (Reference) First | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 20
  Male | 7 | 13 | 20
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 10 | 13 | 23
  Black | 5 | 3 | 8
  Asian | 4 | 3 | 7
  Hispanic | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Trandolapril: Trandolapril 4 mg Tablet (test) dosed in either period
- Mavik®: Mavik® 4 mg Tablet (reference) dosed in either period
Arm/Group | Trandolapril | Mavik®
Number analyzed (Participants) | 37 | 37
pg/mL | 4559.54 (2269.88) | 4872.59 (2218.00)
Statistical Analysis 1: Comparison: Trandolapril vs Mavik®; Test type: Non-Inferiority or Equivalence — Using GLM procedures in SAS, analysis of variance (ANOVA)was performed on log-transformed AUC0-t, AUC0-inf and Cmax at the significance level of 0.05; Ratio of Least Squares Means = 93.26, 90% CI [83.39 to 104.31] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Trandolapril | Mavik®
Number analyzed (Participants) | 37 | 37
pg*h/mL | 4868.37 (2340.05) | 4826.71 (2022.13)
Statistical Analysis 1: Comparison: Trandolapril vs Mavik®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means = 100.35, 90% CI [92.08 to 109.36] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Trandolapril | Mavik®
Number analyzed (Participants) | 37 | 37
pg*h/mL | 4609.82 (2178.05) | 4612.53 (1897.96)
Statistical Analysis 1: Comparison: Trandolapril vs Mavik®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means = 99.17, 90% CI [92.71 to 106.08] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

4. Secondary Outcome: Cmax - Trandolaprilat
Description: Informational Purposes Only
Time Frame: Blood samples collected over 72 hour period
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Trandolapril | Mavik®
Number analyzed (Participants) | 37 | 37
pg/mL | 6682.74 (2005.26) | 6526.16 (1961.47)
Statistical Analysis 1: Comparison: Trandolapril vs Mavik®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means = 102.93, 90% CI [99.80 to 106.15] — Informational Purposes Only

5. Secondary Outcome: AUC0-inf - Trandolaprilat
Description: Informational Purposes Only
Time Frame: Blood samples collected over 72 hour period
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Trandolapril | Mavik®
Number analyzed (Participants) | 37 | 37
pg*h/mL | 138305.28 (25043.67) | 138925.03 (29142.49)
Statistical Analysis 1: Comparison: Trandolapril vs Mavik®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means = 100.24, 90% CI [98.11 to 102.43] — Informational Purposes Only

6. Secondary Outcome: AUC0-t - Trandolaprilat
Description: Informational Purposes Only
Time Frame: Blood samples collected over 72 hour period
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Trandolapril | Mavik®
Number analyzed (Participants) | 37 | 37
pg*h/mL | 111204.01 (18419.42) | 111685.36 (20122.99)
Statistical Analysis 1: Comparison: Trandolapril vs Mavik®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means = 100.10, 90% CI [98.12 to 102.12] — Informational Purposes Only

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.